CLINICAL TRIAL: NCT03168139
Title: A Two-part, Open-label Phase 1/2 Study to Evaluate Pharmacodynamic Effects and Safety of Olaptesed Pegol Monotherapy and Safety and Efficacy of Olaptesed Pegol / Pembrolizumab Combination Therapy in Metastatic Colorectal and Pancreatic Cancer
Brief Title: Olaptesed (NOX-A12) Alone and in Combination With Pembrolizumab in Colorectal and Pancreatic Cancer
Acronym: Keynote-559
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TME Pharma AG (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNOXA12C601; 2016-003657-15 (EudraCT Number); Keynote-559 (Other: NOXXON Pharma/Merck Sharp & Dohme Corp.)
Record Dates: First submitted 2017-05-19; First posted 2017-05-30 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Metastatic Colorectal Cancer; Metastatic Pancreatic Cancer
Keywords: Metastatic colorectal cancer; Metastatic pancreatic cancer; NOX-A12; Olaptesed pegol; Spiegelmer; Pembrolizumab; PD-1 inhibitor; Stromal cell-derived factor-1 (SDF-1); CXCL12; Tumor microenvironment; Immunotherapy; Checkpoint inhibition
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms | interventions — NOX-A12; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olaptesed pegol + Pembrolizumab (Experimental)
  Interventions: Drug: Olaptesed pegol - Monotherapy; Drug: Olaptesed pegol + Pembrolizumab - Combination Therapy

INTERVENTIONS:
Drug: Olaptesed pegol - Monotherapy — Monotherapy (MT) period:
  Treatment with 300 mg olaptesed pegol only, weekly on MT D1 and MT D4 for up to 2 weeks
  Other Names: NOX-A12
Drug: Olaptesed pegol + Pembrolizumab - Combination Therapy — Combination therapy (CT) period:
  Treatment with 300 mg olaptesed pegol in combination with 200 mg pembrolizumab every three weeks (Q3W) until progressive disease or limiting toxicity, for a maximum of 24 months in total
  Other Names: NOX-A12, Keytruda, MK-3475

SUMMARY:
The purpose of this study is to show that the type, number and/or distribution of tumor metastases infiltrating immune cells such as cytotoxic T cells and/or the cytokine signature in the tumor metastases can be modulated by treatment with olaptesed pegol and to explore safety, tolerability and efficacy of olaptesed pegol in combination with pembrolizumab as a basis for subsequent studies in combination with immunotherapies, in particular checkpoint inhibitors.

DETAILED DESCRIPTION:
Olaptesed pegol (NOX-A12) targets a key chemokine in the tumor microenvironment, CXCL12, which is naturally involved in the homeostasis of blood and immune cells. In cancer, CXCL12 acts as a communication bridge between tumor cells and their environment. In particular, it confers resistance to checkpoint inhibitors through T-cell exclusion in preclinical models. The hypothesis is that inactivation of CXCL12 by olaptesed pegol induces changes in the tumor microenvironment of patients with colorectal and pancreatic cancer which render the tumors more susceptible to immuno-oncological approaches such as checkpoint inhibition.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age ≥18 years
3. a) Male or female patient with a history of treated metastatic stage IV colorectal cancer with liver metastases of the primary colorectal cancer after two or more lines of prior treatment OR b) Male or female patient with a history of treated metastatic stage IV pancreatic ductal adenocarcinoma with liver metastases of the primary pancreatic cancer after one or more lines of prior treatment
4. Histologically or cytologically confirmed diagnosis of colorectal or pancreatic ductal cancer with liver metastasis
5. Measurable disease based on RECIST 1.1 as determined by the site study team
6. Expected survival of at least three months
7. Patient with liver metastasi(e)s amenable to repeated biopsies
8. Patient agreeing to repeated biopsies of metastases
9. Karnofsky performance status ≥80 %
10. a) Colorectal cancer patients that have received current standard treatment options (progression or intolerance to oxaliplatin, irinotecan, 5-fluorouracil and trifluridine/tipiracil with or without treatment combinations of cetuximab and/or bevacizumab, or ramucirumab or panitumumab, or regorafenib, including monotherapies with any of these options) OR b) Pancreatic cancer patients that have received current treatment options (progression or intolerance to combination therapies with oxaliplatinum, irinotecan, 5-fluorouracil, gemcitabine, nab-paclitaxel or erlotinib, including monotherapies with any of these options)
11. No chemotherapy treatment within the last three weeks prior to study MT Day 1
12. Resolution of toxic effect(s) of the most recent prior chemotherapy to levels deemed appropriate by the investigator; if patients have received major surgery, they must have recovered from the toxicity and/or complications from the intervention
13. The following laboratory parameters should be within the ranges specified:

    * Hemoglobin (Hb) ≥ 8.0 g/dL
    * Absolute neutrophil count (ANC) ≥ 1,000/mm³ (≥ 1.0 x 10^9/L)
    * Platelets ≥ 100,000/mm³ (≥ 100 x 10^9/L)
    * Creatinine ≤ 1.5 x ULN or glomerular filtration rate ≥ 60 mL/min/1.73m²
    * Total bilirubin ≤ 1.5 x ULN (upper limit normal)
    * ALT (alanine transaminase) ≤ 5 x ULN
    * AST (aspartate transaminase) ≤ 5 x ULN
    * INR (International Normalized Ratio) or PT (Prothrombin Time) ≤ 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
    * aPTT (Activated Partial Thromboplastin Time) ≤ 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
14. Female patients of child-bearing potential must have a negative urine or serum pregnancy test within 28 days prior to randomization. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Patients must agree to use an effective method of contraception or be abstinent during and for 120 days following last dose of drug (more frequent pregnancy tests may be conducted if required per local regulations)
15. Male patients must use an effective barrier method of contraception during study and for 120 days following the last dose if sexually active with a FCBP

Exclusion Criteria:

1. Inability to personally provide written informed consent or to understand and collaborate throughout the study
2. Inability or unwillingness to comply with study requirements
3. Patients with metastatic lesions suitable for resection
4. Patients with metastatic cancer that have a drastic clinical progression (e.g. from Karnofsky performance 100% to 70%) within the last six weeks before screening
5. Participation in any clinical research study with administration of an investigational drug or therapy within 30 days prior to enrolment in the study
6. Use of any investigational or non-registered product (drug or vaccine) other than the study treatment
7. Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or if the patient has previously participated in pembrolizumab clinical studies
8. Prior radiation therapy of tumor/metastases
9. Diagnosis of immunodeficiency or requiring concomitant chronic treatment with systemic corticosteroids or any other immunosuppressive agents within 7 days prior to the first dose of study treatment; the use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor
10. Intake of immunomodulatory medication (Type 1 interferons)
11. Prior anti-cancer monoclonal antibody (mAb) within 2 weeks prior to study MT Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to such agents administered more than 2 weeks earlier
12. Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study MT Day 1 or no recovery (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent
13. Prior transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including G-CSF, GM-CSF or recombinant erythropoietin) within 4 weeks prior to study MT Day 1
14. Live vaccine within 30 days prior to the first dose of study treatment
15. Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
16. History of interstitial lung disease
17. History of (non-infectious) pneumonitis that required steroids or current pneumonitis
18. History of anaphylaxis or severe drug hypersensitivity reactions
19. Active infection requiring systemic therapy
20. Known to be positive for Human Immunodeficiency Virus (HIV) or other chronic infections (HBV, HCV) or with another confirmed or suspected immunosuppressive or immunodeficient condition
21. Concurrent chronic severe medical problems (heart failure, uncontrolled diabetes, bleeding disorder etc.), unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk
22. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
23. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
24. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator, is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment
25. Women of childbearing potential: refusal or inability to use effective means of contraception
26. Contra-indication or known hypersensitivity to olaptesed pegol, polyethylene glycol, pembrolizumab or further ingredients to the investigational medicinal products
27. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
28. Previous enrolment in this clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Monotherapy: Pharmacodynamics | up to 14 days
  Evaluation of changes within the tumor microenvironment induced by CXCL12 inhibition with olaptesed pegol by comparing pre- and post-treatment biopsy specimens
Combination Therapy: Safety - adverse events, vital signs, ECG, hematology & safety laboratory | up to 24 months
  Safety and tolerability of olaptesed pegol in combination with pembrolizumab will be evaluated by assessing adverse events, vital signs (pulse rate, blood pressure), 12-lead ECG, hematology (full blood count including platelets and differential count), safety laboratory including thyroid function tests

SECONDARY OUTCOMES:
Monotherapy: Safety | up to 14 days
  Assessment of safety and tolerability of olaptesed pegol in patients with metastatic (stage IV) colorectal and pancreatic cancer (adverse events, vital signs (pulse rate, blood pressure), 12-lead ECG, hematology (full blood count including platelets and differential count), safety laboratory)
Monotherapy: Pharmacodynamics | up to 14 days
  Investigation of changes in the cytokine/chemokine signature within the tumor microenvironment and in the peripheral blood induced by CXCL12 inhibition with olaptesed pegol by comparing the pre- and post-treatment samples
Combination Therapy: Disease control rate (DCR) | up to 24 months
  DCR will be calculated as the proportion of patients with best overall response to treatment with olaptesed pegol in combination with pembrolizumab of complete response (CR), partial response (PR) or stable disease (SD).
  Treatment responses will be assessed according to the current guidelines of the RECIST 1.1 and irRECIST.
Combination Therapy: Efficacy - time to event analyses | up to 24 months
  Efficacy of treatment with olaptesed pegol in combination with pembrolizumab (PFS and OS)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationales Centrum für Tumorerkrankungen (NCT) Heidelberg, Heidelberg, Germany